CLINICAL TRIAL: NCT00002717
Title: A Phase III Randomized Trial of Cisplatin (NSC #119875) With Paclitaxel (NSC #125973) Administered by Either 24 Hour Infusion or 96 Hour Infusion in Patients With Selected Stage III and Stage IV Epithelial Ovarian Cancer and Primary Peritoneal Carcinoma
Brief Title: Paclitaxel and Cisplatin in Treating Patients With Stage III or Stage IV Ovarian Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064554; GOG-0162
Record Dates: First submitted 1999-11-01; First posted 2004-06-22 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2010-01

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective for ovarian or peritoneal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of paclitaxel plus cisplatin in treating patients who have residual disease after surgery to remove stage III or stage IV ovarian cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare progression free and overall survival and frequency of response in patients with suboptimal stage III or IV ovarian epithelial cancer or primary peritoneal cancer treated with a 24 hour vs 96 hour infusion of paclitaxel (TAX) followed by cisplatin. II. Determine the incidence and severity of adverse events, including catheter complications and drug toxicity, for the 96 hour infusion of TAX. III. Compare the relationship between plasma TAX concentrations, toxicity, and response to both infusion schedules in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and measurable disease (yes vs no). Patients are randomized into one of two treatment arms. Arm I: Patients receive paclitaxel IV continuously over 24 hours followed by cisplatin IV over 2 hours. Arm II: Patients receive paclitaxel IV continuously over 96 hours followed by cisplatin IV over 2 hours. Treatment repeats every 3 weeks for 6 courses.

PROJECTED ACCRUAL: A total of 324 patients will be accrued for this study over 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary ovarian epithelial cancer or primary peritoneal cancer Suboptimal residual disease within 6 weeks of laparotomy with maximum resection Stage III residual retroperitoneal disease greater than 1 cm and no greater than 1 cm residual intraperitoneal disease OR Stage IV disease The following histologies are eligible: Serous adenocarcinoma Malignant Brenner's tumor Mucinous adenocarcinoma Endometrioid adenocarcinoma Undifferentiated carcinoma Clear cell adenocarcinoma Mixed epithelial carcinoma Transitional cell carcinoma Adenocarcinoma not otherwise specified Measurable disease not required Cytologic confirmation of malignant pleural effusion required if sole basis of entry No borderline (low malignant potential) carcinoma No unclassified ovarian cancer, i.e., thought to be of ovarian origin but unexplored or unable to verify tumor arising from ovarian stroma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Hematopoietic: WBC at least 3,000/mm3 Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal AST, ALT, and GGT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal LDH no greater than 3 times normal No acute hepatitis Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No history of congestive heart failure No history of unstable angina No myocardial infarction within 6 months Other: No severe infection, including septicemia No severe gastrointestinal bleeding No history of second malignancy within 5 years except nonmelanomatous skin cancer Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics No more than 6 weeks since staging laparotomy and primary cytoreductive surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 1996-03; Primary Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (52):
- United States (52):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Background] Farley JH, Tian C, Rose GS, Brown CL, Birrer M, Maxwell GL. Race does not impact outcome for advanced ovarian cancer patients treated with cisplatin/paclitaxel: an analysis of Gynecologic Oncology Group trials. Cancer. 2009 Sep 15;115(18):4210-7. doi: 10.1002/cncr.24482. PMID 19536873
- [Background] Zorn KK, Tian C, McGuire WP, Hoskins WJ, Markman M, Muggia FM, Rose PG, Ozols RF, Spriggs D, Armstrong DK. The prognostic value of pretreatment CA 125 in patients with advanced ovarian carcinoma: a Gynecologic Oncology Group study. Cancer. 2009 Mar 1;115(5):1028-35. doi: 10.1002/cncr.24084. PMID 19156927
- [Background] Winter WE 3rd, Maxwell GL, Tian C, Sundborg MJ, Rose GS, Rose PG, Rubin SC, Muggia F, McGuire WP; Gynecologic Oncology Group. Tumor residual after surgical cytoreduction in prediction of clinical outcome in stage IV epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2008 Jan 1;26(1):83-9. doi: 10.1200/JCO.2007.13.1953. Epub 2007 Nov 19. PMID 18025437
- [Result] Spriggs DR, Brady MF, Vaccarello L, Clarke-Pearson DL, Burger RA, Mannel R, Boggess JF, Lee RB, Hanly M. Phase III randomized trial of intravenous cisplatin plus a 24- or 96-hour infusion of paclitaxel in epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Oct 1;25(28):4466-71. doi: 10.1200/JCO.2006.10.3846. PMID 17906207
- [Result] Spriggs DR, Brady M, Rubin S, et al.: A phase III randomized trial of cisplatin and paclitaxel administered by either 24 hour or 96 hour infusion in patients with selected stage III or stage IV epithelial ovarian cancer (GOG162). [Abstract] J Clin Oncol 22 (Suppl 14): A-5004, 450s, 2004.
- [Derived] Rose PG, Java JJ, Salani R, Geller MA, Secord AA, Tewari KS, Bender DP, Mutch DG, Friedlander ML, Van Le L, Method MW, Hamilton CA, Lee RB, Wenham RM, Guntupalli SR, Markman M, Muggia FM, Armstrong DK, Bookman MA, Burger RA, Copeland LJ. Nomogram for Predicting Individual Survival After Recurrence of Advanced-Stage, High-Grade Ovarian Carcinoma. Obstet Gynecol. 2019 Feb;133(2):245-254. doi: 10.1097/AOG.0000000000003086. PMID 30633128